CLINICAL TRIAL: NCT02282475
Title: Role of Liver and Visceral Fat in Glucose and Lipid Metabolism During Pregnancy
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01DK098707-01A1 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2014-11-04 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Pregnancy; Gestational Diabetes; Obesity; Liver Fat
MeSH Terms: conditions — Diabetes, Gestational; Obesity; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort study of pregnant women: Participants will complete the following at 12-16 weeks gestation and again at 32-36 weeks gestation:
  1. Fasting glucose, insulin and insulin sensitivity testing;
  2. Blood tests for cholesterol and fatty acids, liver function, inflammation, and markers of metabolism;
  3. Measurements of body fat using air displacement technology and MRI;
  4. Ultrasound to measure placental blood flow, visceral fat thickness (12-16 weeks only) and to estimate fetal weight (32-36 weeks only);
  5. 24 hour diet recalls
  6. Questionaires regarding activity level
- Case-control study Gestational Diabetes: Participants diagnosed with gestational diabetes (cases) and without gestational diabetes (controls) will complete the following at 32-36 weeks gestation:
  1. Fasting glucose, insulin and insulin sensitivity testing;
  2. Blood tests for cholesterol and fatty acids, liver function, inflammation, and markers of metabolism;
  3. Measurements of body fat by using air displacement technology and MRI;
  4. Ultrasound to measure placental blood flow and to estimate fetal weight;
  5. 24 hour diet recalls
  6. Questionaires regarding activity level

SUMMARY:
Obesity, increased abdominal fat, fat stored in the liver, and insulin resistance may all be associated with adverse maternal and fetal pregnancy outcomes. This study will examine how fat storage changes during pregnancy; and if how the body stores fat impacts one's ability to metabolize glucose (sugar) during pregnancy.

DETAILED DESCRIPTION:
This study aims to serially evaluate liver and visceral fat stores during pregnancy and their relationship with glucose and lipid metabolism, placental function, and newborn size. To do this we will conduct both a prospective cohort study of pregnant women without pre-gestational or early gestational diabetes assessed at both 12-16 weeks gestation and at 32-36 weeks gestation and a case-control study of women with normal and impaired glucose tolerance in the early third trimester. Physical assessments will be performed by the Oregon Health and Science University bio-nutrition unit and will include the use of magnetic resonance imaging, ultrasound, and blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and enrolled members of Kaiser

Exclusion Criteria:

* Women with multiples pregnancy; history of: cardiovascular disease, bariatric surgery, anemia, chronic hypertension or renal disease.
* Non-English speaker

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women ages 18-40 years and actively enrolled in Kaiser Permanente Northwest (KPNW).
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Assess visceral adipose fat and intrahepatic lipid stores change during pregnancy | 12-16 weeks and 32-36 weeks gestation
  We will compare visceral adipose fat and intrahepatic lipid levels in early pregnancy (12-16 weeks gestation) to late pregnancy (32-36 weeks gestation). This will done by comparing changes in accumulation of fat in the visceral adipose tissue, changes in intrahepatic lipid values and changes in total body fat in early and late pregnancy. We will be collecting body composition measurements and utilizing ultrasound and Magnetic Resonance Imaging.

SECONDARY OUTCOMES:
Compare glucose tolerance in pregnant women with gestational diabetes to those with normal glucose tolerance | 34 weeks gestation
  We will use a matched case-control design with matching for body mass index to compare intrahepatic lipid, visceral adipose tissue, total body fat, and insulin sensitivity among women with gestational diabetes and normal glucose tolerance, as measured at 32-36 weeks gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Vesco, MD, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: No